CLINICAL TRIAL: NCT06672159
Title: A Randomized Controlled Trial on Early Double External Sequential Defibrillation in Out of Hospital Cardiac Arrest
Brief Title: Initial Double Sequential External Defibrillation in Out of Hospital Cardiac Arrest
Acronym: DUALDEFIB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian Air Ambulance Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 724951
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrest; Out-Of-Hospital Cardiac Arrest; Ventricular Fibrillation
Keywords: Double defibrillation; Cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation

STUDY DESIGN:
Intervention Model Description: All included ambulance stations will perform one of the two procedures for six months followed by a crossover for six months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double sequential external defibrillation (Experimental): Patient will receive first shock using two defibrillators. All other aspects of resuscitation in accordance to existing guidelines.
  Interventions: Device: Two defibrillators
- Standard treatment (Active Comparator): Standard treatment in accordance to existing Advanced Cardiopulmonary Resuscitation-guidelines using one defibrillator in anterior-lateral placement.
  Interventions: Device: One defibrillator

INTERVENTIONS:
Device: Two defibrillators — DSED procedure consists of pads placed in anterior-lateral position, and in anterior-posterior position. Defibrillations will be given in rapid sequence, less than a second apart. All other aspects of resuscitation in accordance to existing guidelines.
  Arms: Double sequential external defibrillation
Device: One defibrillator — Standard OHCA treatment according to existing guidelines.
  Arms: Standard treatment

SUMMARY:
Double Sequential External Defibrillation (DSED) represents an alternative treatment of refractory ventricular fibrillation (rVF) in out-of-hospital cardiac arrest (OHCA). The procedure consists of two defibrillators that administer shocks at the same time.

Currently, the procedure is not initiated before at least three failed attempts with one defibrillator. This can delay the potential benefits of establishing DSED earlier in the treatment. Studies have shown that early defibrillation is crucial for survival in OHCA patients, and in 2022, a clinical trial showed that survival in patients treated with DSED was higher compared to standard treatment.

The effect of initiating OHCA treatment is unknown. The DUALDEFIB trial seeks to investigate if treating OHCA patients with DSED as an initial treatment will increase survival and provide improved neurological outcome.

DETAILED DESCRIPTION:
The project is investigator-initiated, prospective, two-group randomized controlled trial (RCT). Prior to the RCT, a pilot feasibility trial of 3-4 months will be performed, including three ambulance bases in mid-Norway. All OHCA patients will be included until validity and feasibility of the study is accomplished. The pilot study will be followed by the RCT.

Outcome measurements in the RCT are aimed to be the same as in the pilot study. Ambulance bases will be randomized to either DSED or standard procedure for six months before crossover with the other treatment for six months.

Ambulances included in the project will carry two defibrillators. Both defibrillators will be established for initial defibrillation with DSED in OHCA patients. The pads are placed in anterior-lateral position (standard placement) and anterior-posterior position (over sternum and beneath left scapula). Shocks are administered in rapid succession with less than one second apart. All other treatment will be according to existing guidelines.

The included patients are OHCA patients with age over 18 years presenting with a shockable rhythm. Excluded patients are patients with obvious or suspected pregnancy, incarcerated patients or patients with no-resuscitation order. The patients that meet the inclusion criteria will be registered by the ambulance personnel through a secure webpage.

Primary outcome is survival to hospital admission.

Secondary outcomes are survival to hospital discharge, 30 days, 90 days and 1 year survival, in addition to neurological status.

Patients from the pilot will be included in the RCT intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with out of hospital cardiac arrest presenting with a shockable rhythm

Exclusion Criteria:

* Age below 18 years
* Obvious or suspected pregnancy
* Incarcerated patients
* Preexisting do-not-resuscitate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that survive to hospital admission. | 24 hours
  Number of patients arriving with ROSC in hospital emergency facility.

SECONDARY OUTCOMES:
Proportion of patients that survive for 30 days | 30 days
  Number of patients that have survived OHCA incident after 30 days.
Review of 30 day neurological status. | 30 days
  Modified Rankin Scale (1 No significant disability - 5 Severe disability) defines neurological outcome of OHCA.
Proportion of patients that survive for 90 days | 90 days
  Number of patients that have survived OHCA incident after 90 days.
Review 90 day neurological status. | 90 days
  Modified Rankin Scale (1 No significant disability - 5 Severe disability) defines neurological outcome of OHCA.
Proportion of patients that survive for one year. | 365 days
  Number of patients that have survived OHCA incident after 365 days.

OTHER OUTCOMES:
Incidence of patient-related adverse effects. | 365 days
  Measure/obtain information regarding adverse effects experience by patient using DSED procedure.
Incidence of malfunction of defibrillator. | 365 days
  Assess information regarding occurrence of defibrillator damage after DSED procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Karlsen, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol, statistical analysis plan, information letter for consent and other trial documents will be published open access. The clinical study report and statistical analysis report will also be made openly available but may be altered to hide information that may lead to identification of individual study participants.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol and ICF will be available before study start. SAP will be available before first interim analysis.
Access Criteria: Individual level data will be made available to sponsor institutions. Access will be controlled by a data processor agreement between the partner and funder. De-identified individual level data collected during the trial, will be made available on request to researchers from other scientific institutions by approval of the project management to ensure that usage is compliant with privacy and consent requirements as well as conditions for attribution and usage. Data sharing with editors or peer-reviewers of scientific journals, conferences or the like will not require additional consent or data access agreement with sponsor, as such data will not be shared onward or used beyond reviewing this trial.
  After data sharing, the sponsor must be acknowledged in any publication resulting from the shared data. For closer collaboration attribution based on the Vancouver Convention will apply.

DOCUMENTS (1):
  • Study Protocol (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT06672159/Prot_000.pdf